CLINICAL TRIAL: NCT03697395
Title: Advanced Immunoclinical Phenotyping of Rejection in Lung Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Y. Michael Shim, MD, Associate Professor of Medicine and Medical Imaging, University of Virginia
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20987; Ithriv (Other: National Institute of Health)
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Chronic Rejection of Lung Transplant

STUDY DESIGN:
Intervention Model Description: Part 1-blood and bronch samples will be collected from subjects already undergoing procedures Part 2-blood, bronch samples and MRI will be performed on subject
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Lung transplant recipient without MRI imaging — Patients who received lung transplant and undergoing surveillance follow-up at 1, 3, 6, 12, 24 months after the date of lung transplant, but without consenting to be evaluated by hyperbolized gas MRI. Bronchoscopy sampling will be performed per usual lung transplant team protocol.
  Other Names: Routine Lung Transplant Surveillance
Drug: Lung transplant recipient with MRI imaging — Patients who received lung transplant and undergoing surveillance follow-up at 1, 3, 6, 12, 24 months after the date of lung transplant and with consenting to be evaluated by hyperbolized has MRI. Bronchoscopy sampling will be guided by the results of the hyper polarized gas MRI, different from the usual lung transplant team protocol. Administration of hyper polarized gas MRI is under FDA regulation by IND #129769 (PI, Yun Michael Shim, MD)
  Other Names: Lung Transplant Surveillance with hyper polarized gas MRI

SUMMARY:
Chronic allograft rejection of the transplanted lung (CLAD) is a major health issue in patients after lung transplant. This study is a registry-forming study with concurrent tissue banking from surveillance bronchoscopy in addition to extra tissue sampling of blood and urine. Patients will be characterized by usual clinical phenotyping and the latest imaging methods so that diseased condition underlying CLAD can be better understood.

DETAILED DESCRIPTION:
Chronic allograft rejection of the transplanted lung (CLAD) is a major health issue that lead to almost 50% mortality within 5 years from the time of lung transplant. In the past CLAD was exclusively occurring in small airways causing a condition called "Bronchiolitis Obliteran Syndrome" (BOS). However, recently many have observed restrictive changes in lung physiology with or without parenchymal abnormalities. This new CLAD is called RAS or RCLAD. What is also concerning is that RAS is thought to be associated with disproportionally high morbidity and mortality. This clinical trial intends to create a registry of patients who completed lung transplant and who are undergoing routine surveillance bronchoscopy. A subgroup of patients will be characterized by hyper polarized gas magnetic resonance image to enhance detection of CLAD, and to be correlated between the MRI imaging results and clinical/biochemical results. This study is anticipated to advance our understanding of CLAD which is currently inevitably fatal outcome among patients after lung transplant.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who successfully underwent lung transplant at the University of Virginia.
2. Followed by medical lung transplant team for post-lung transplant rejection surveillance program at the University of Virginia.
3. Subjects with co -morbid illnesses such as neurologic, liver and or kidney or GI tract disease/ dysfunction are not excluded
4. Clinically stable to undergo MRI Imaging

Exclusion Criteria:

1. Continuous oxygen use at home if decided to consent for MRI imaging
2. Blood oxygen saturation of less than 92%as measured by pulse oximetry on the day of imaging if decided to consent for MRI imaging.
3. Forced Expiratory Volume in 1 second (FEV1) percent predicted less than 25% if decided to consent for MRI imaging.
4. Pregnancy or lactation if decided to consent for MRI imaging.
5. Claustrophobia, inner ear implants, aneurysm or other surgical clips, metal foreign bodies in eye, pacemaker or other contraindication to MR scanning. Subjects with any implanted device that cannot be verified as MRI compliant will be excluded if decided to consent for MRI imaging.
6. Chest circumference greater than that of the xenon MR and/or helium coil. The circumference of the coil is approximately 42 inches if decided to consent for MRI imaging.
7. History of congenital cardiac disease, chronic renal failure, or cirrhosis if decided to consent for MRI imaging.
8. Inability to understand simple instructions or to hold still for approximately 10 seconds if decided to consent for MRI imaging.
9. History of respiratory infection within 2 weeks prior to the MR scan if decided to consent for MRI imaging.
10. History of MI, stroke and/or poorly controlled hypertension if decided to consent for MRI imaging.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful collection of all samples as proposed. | 24 months after the date of lung transplant surgery
  Completion of surveillance bronchoscopy and other tissue collection at planned surveillance (24 months after the date of lung transplant surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Yun M Shim, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No